CLINICAL TRIAL: NCT04650100
Title: Analgesic Effectiveness of PENG Block in Programmed Hip Arthroplasty Surgery
Acronym: THAPeng
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RC31/20/0227; 2020-A01887-32 (Other: ID-RCB)
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Pain
Keywords: Total hip arthroplasty; PENG bloc; local anaesthetics infiltration; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG group (Experimental): For the PENG group, the ultrasound-guided PENG block (20 ml of Ropivacaine 4.75 mg/ml) is performed before the surgery.
  Interventions: Procedure: ultrasound-guided PENG bloc realized before surgery
- Control group (No Intervention): No additional intervention, only standard care

INTERVENTIONS:
Procedure: ultrasound-guided PENG bloc realized before surgery — ultrasound-guided PENG block realized before surgery. The PENG block, described by Giron-Arebgi is made in the supine position. The ultrasound probe used is a 5 MHz high frequency linear probe placed parallel to the line delimited by the anterior-inferior iliac spine (lateral) and the pubis (medial). The needle used is an 80 mm, 22G, needle inserted in the ultrasound plane. The slow and fractioned injection of 20 ml of Ropivacaine 4.75 mg/ml is performed in the fascia between the psoas tendon and the iliopubic eminence under ultrasound guidance.
  Arms: PENG group

SUMMARY:
The intra- and peri-articular infiltration of local anaesthetics realized at the end of total hip arthroplasty surgeries is an effective analgesic technique, but it can be insufficient to manage the possibly intense postoperative pain. Regional anaesthesia (RA) like the recently described pericapsular nerve group (PENG) block could provide additional analgesic benefit in this setting.

Investigators main objective is to demonstrate the analgesic benefits (postoperative pain score and morphine consumption) of the PENG block when added to intra- and peri-articular infiltration of local anaesthetic following total hip arthroplasty. Investigators make the assumption that i) the PENG bloc could reduce the postoperative 24 first hours morphine consumption by 30%, ii) the PENG block could spare the motor function of the quadriceps and adductor muscles, and iii) the PENG bloc could be well tolerated allowing a high level of patient satisfaction.

DETAILED DESCRIPTION:
A recent study has revealed a region of pericapsular terminal branches of the femoral nerve and the obturator nerve accessible to ultrasound-guided regional anaesthesia. This technique, also called the PENG block, has recently been described with a substantial benefit on pain at rest and induced by mobilization in cases series of patients undergoing hip fracture surgery. To investigators knowledge, no randomized data concerning the analgesic efficacy of the PENG block has been published in the setting of elective total hip arthroplasty.

The PENG block would allow a significant analgesic contribution when added to intra- and peri-articular infiltration of local anaesthetics while being well tolerated with few undesirable effects. Moreover, the PENG block could spare the motor function of the quadriceps and adductor muscles allowing enhanced recovery after surgery

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for total hip arthroplasty surgery under general anaesthesia
* Affiliated of a social security scheme
* Having signed the written informed consent

Exclusion Criteria:

* Total hip arthroplasty revision surgery
* Refusal of the patient to participate
* Existence of major spontaneous or acquired haemostasis disorders
* Infection at the puncture site
* Allergy to local anaesthetics
* Pregnancy or breast-feeding
* Patients under the protection of adults (guardianship, curatorship or protection of justice)
* Patients whose cognitive state does not allow assessment by the scales used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Cumulated postoperative morphine consumption 24 hours after surgery | 24 hours
  calcul of Cumulated postoperative morphine consumption 24 hours after surgery

SECONDARY OUTCOMES:
Cumulated postoperative morphine consumption in the post anaesthesia care unit (PACU) | Hour 1
  Cumulated postoperative morphine consumption in the post anaesthesia care unit (PACU)
Cumulated postoperative morphine consumption 48 hours after surgery | Hour 48
  Cumulated postoperative morphine consumption 48 hours after surgery
Evaluation of pain in the PACU | Hour 1
  Evaluation of pain using a simple numeric rating scale (NRS from 0 to 10) in the PACU
Evaluation of pain 24 hours after surgery | Hour 24
  Evaluation of pain using a simple numeric rating scale (NRS from 0 to 10) 24 hours after surgery
Evaluation of pain 48 hours after surgery | Hour 48
  Evaluation of pain using a simple numeric rating scale (NRS from 0 to 10) 48 hours after surgery
Evaluation of the pain potentially induced by the realization of the PENG block | Hour 0
  Evaluation of the pain potentially induced by the realization of the PENG block with Likert scale from 1 to 5, 1 is for no pain, 5 is for the worse pain
Evaluation of adverse effects associated with the PENG block | Hour 0
  Evaluation of adverse effects associated with the PENG block
Evaluation of adverse effects associated with the PENG block | Hour 1
  Evaluation of adverse effects associated with the PENG block
Evaluation of adverse effects associated with the PENG block | Hour 24
  Evaluation of adverse effects associated with the PENG block
Evaluation of adverse effects associated with the PENG block | Hour 48
  Evaluation of adverse effects associated with the PENG block
Evaluation of adverse effects associated with the use of morphine | Hour 0
  Evaluation of adverse effects associated with the use of morphine
Evaluation of adverse effects associated with the use of morphine | Hour 1
  Evaluation of adverse effects associated with the use of morphine
Evaluation of adverse effects associated with the use of morphine | Hour 24
  Evaluation of adverse effects associated with the use of morphine
Evaluation of adverse effects associated with the use of morphine | Hour 48
  Evaluation of adverse effects associated with the use of morphine
Evaluation of the patients' satisfaction | Hour 24
  Evaluation of the patients' satisfaction by the EVAN-LR score realized 24 hours after surgery. EVAN-LR is a scale assessing perioperative patient's satisfaction with Loco Regional anaesthesia
Evaluation of the adductor muscles weakness | Hour 24
  Evaluation of the adductor muscles weakness by a thigh adduction test performed 24 hours after surgery
Evaluation of the quadricipital muscles weakness | Hour 24
  Evaluation of the quadricipital muscles weakness by a Timed to Up and Go Test performed 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: FERRE Fabrice, PH, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ferre F, Rey J, Bosch L, Menut R, Ferrier A, Ba C, Halimi C, Collinson I, Tissot B, Labaste F, Reina N, Minville V. Pericapsular nerve group (PENG) block combined with local infiltration analgesia is not superior to local infiltration analgesia for the management of postoperative pain after primary elective total hip arthroplasty: A prospective, randomized, controlled, single-blind trial. Heliyon. 2024 Jun 27;10(13):e33766. doi: 10.1016/j.heliyon.2024.e33766. eCollection 2024 Jul 15. PMID 39071707